CLINICAL TRIAL: NCT06495034
Title: A Randomized Controlled Study on Early Intervention of Airwave Compression Therapy to Prevent Breast Cancer-related Upper Limb Lymphedema
Brief Title: Airwave Compression Therapy to Prevent Breast Cancer-related Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shantou Central Hospital (Other)
Responsible Party: Principal Investigator, Si-Qi Qiu, Principal Investigator, Shantou Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ShantouCH003
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: breast cancer-related lymphedema; airwave compression therapy; quality of life
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): standard care: health education and routine functional exercise
  Interventions: Other: standard care: health education and routine functional exercise
- experimental group (Experimental): 1. standard care: health education and routine functional exercise;
  2. airwave compression therapy
  Interventions: Device: airwave compression therapy; Other: standard care: health education and routine functional exercise

INTERVENTIONS:
Device: airwave compression therapy — Airwave compression therapy was given to patients after breast cancer surgery to treat the ipsilateral upper limb
  Other Names: Airwave pressure therapy，intermittent pneumatic compression pump，IPC
  Arms: experimental group
Other: standard care: health education and routine functional exercise — standard care: health education and routine functional exercise

SUMMARY:
This study aims to explore the effectiveness of early intervention of airwave compression therapy to prevent the occurrence of postoperative breast cancer-related lymphedema(BCRL).

DETAILED DESCRIPTION:
This study aims to explore the effectiveness of early intervention of airwave compression therapy to prevent the occurrence of postoperative breast cancer-related lymphedema (BCRL), hereby improving the quality of life of patients with breast cancer. Furthermore, we will perform exploratory analyses to investigate the predictive values of patient plasma cytokines to the occurrence and development of BCRL.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this clinical trial. Fully understand and be informed about the study and sign an informed consent form (ICF). Willing to follow and able to complete all test procedures;
* Female, ≥18 years old and ≤70 years old at the time of signing the ICF;
* Patients with unilateral breast cancer diagnosed by histopathology or cytology;
* No distant metastasis;
* To undergo unilateral axillary sentinel lymph node biopsy or unilateral axillary lymph node dissection;
* Have not received any treatment for arm lymphedema;
* No lymphangitis and other infections.

Exclusion Criteria:

* Breast malignancy derived from other tumors rather than the primary breast cancer;
* Patients with second primary tumor;
* Contraindication to airwave compression therapy: Acute venous thrombosis; Acute inflammatory skin disease; Erysipelas; Arrhythmia; Pulmonary edema; Unstable hypertension; People with artificial pacemakers; Deep thrombophlebitis;
* Have a history of mental illness or other reasons can not cooperate with treatment;
* Embolism, cardiogenic edema, hepatogenic edema and the history of upper limb trauma and other related complications;
* Patients using any medication that affects fluid or electrolyte balance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of lymphedema | 18 months
  Incidence of lymphedema of ipsilateral upper limb

SECONDARY OUTCOMES:
Symptoms | 18 months
  Questionnaire. The level of subjective symptoms( pain, heaviness, paresthesia) at each time point was recorded with a 0-3 four-point scale questionnaire. 0-3 indicated no symptoms, mild, moderate, and severe, respectively.
Quality of life assessment | 18 months
  FACT-B (V4.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Shantou Central Hospital, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No